CLINICAL TRIAL: NCT06147661
Title: Primary Aesthetic Breast Augmentation: Comparative Study Between Breast Implants and Autograft of Adipose Tissue
Acronym: AMEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8954
Record Dates: First submitted 2023-10-26; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-10

CONDITIONS: Breast Implants
Keywords: Breast Prosthesis; Breast Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of autograft of adipose tissue for aesthetic breast augmentation is increasing year after year. According to the latest meta-analysis of 2016, autograft of adipose tissue in augmentation mastoplasty seems to be a promising method with a satisfactory resorption volume and patient and surgeon satisfaction. However, this technique allows for small to moderate breast augmentation and is therefore not suitable for patients wanting a significant increase.

Breast prostheses allow a significant increase. Numerous studies have shown an improvement in patient satisfaction and quality of life assessed using the BREAST-Q questionnaire.

On the other hand, very few studies have objectively evaluated the satisfaction of patients who have benefited from an autograft of adipose tissue as part of aesthetic breast augmentation. No study has yet compared the satisfaction of patients who have benefited from breast implants or lipofilling.

The aim of this study is to compare the satisfaction of patients who have benefited from breast augmentation by prosthesis or by lipofilling using a remote satisfaction interview.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (age ≥ 18 years)
* having benefited from primary aesthetic breast augmentation at Strasbourg University Hospital between June 27, 2017 and June 27, 2022
* not opposing the reuse of its data for scientific research purposes.

Exclusion Criteria:

* Woman who expressed her opposition to the reuse of her data for scientific research purposes
* Woman with a breast malformation: tuberous breasts or breast asymmetry of more than one cup
* Woman with comprehension difficulties
* Woman under guardianship or curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult woman (age ≥ 18 years) having benefited from primary aesthetic breast augmentation at Strasbourg University Hospital between June 27, 2017 and June 27, 2022
Sampling Method: Non-Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01-22 (Estimated)

PRIMARY OUTCOMES:
Patient woman satisfaction | 1 to 4 years after breast implants
  This satisfaction will be assessed using a remote satisfaction interview

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Plastique, Reconstructrice et Esthétique - CHU de Strasbourg - France, Strasbourg, France